CLINICAL TRIAL: NCT05195359
Title: The Effects of a Personalized Sleep Improvement Smartphone Application From SleepScore Labs: A Single-blinded Randomized Waitlist Controlled Trial
Brief Title: The Effects of a Personalized Sleep Improvement App From SleepScore Labs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Collaborators: SleepScore Labs International LTD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20211202DSDT
Record Dates: First submitted 2021-12-03; First posted 2022-01-19 (Actual); Results first posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Health Behavior
Keywords: Sleep; Smartphone Application; Preventative Health
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: Single-blinded Randomized Waitlist Controlled Trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allocation to Sleep Improvement App (Active Comparator): Participants will be instructed to engage with the Dein Schlaf. Dein Tag. smartphone app, log their behaviors in-app, and track their sleep daily for the duration of the study (12 weeks). Participants will be instructed to start the sleep tracking device via their iOS device before lying down in bed and turning off the lights to go to sleep. In the morning, participants will turn off the sleep tracking device as soon as they wake up and decide to leave the bed. At the three time points (baseline, 6 weeks, and 12 weeks), participants will be instructed to complete online assessments on self-reported sleep quality, health perception, psychosocial factors and sleep-permissive behaviors (i.e., preventative health)
  Interventions: Behavioral: Dein Schlaf. Dein Tag. sleep improvement application powered by SleepScore
- Allocation to Waitlist Control Group (No Intervention): At the three time points (baseline, 6 weeks, and 12 weeks) participants assigned to the wait-list control group will be instructed to complete online assessments on self-reported sleep quality, health perception, psychosocial factors and sleep-permissive behaviors (i.e., preventative health)

INTERVENTIONS:
Behavioral: Dein Schlaf. Dein Tag. sleep improvement application powered by SleepScore — The Dein Schlaf. Dein Tag. application powered by SleepScore is a validated sleep measurement application using sonar technology that also provides evidenced-based sleep advice and sleep education content based on a user's objectively measured nightly sleep data. As participants engage with the app, the Dein Schlaf. Dein Tag. application provides personalized and dynamic sleep content and sleep and circadian rhythm improvement advice based in the principles of sleep hygiene, sleep-circadian science, and cognitive behavioral psychology. Participants will also receive personalized sleep challenges tailored to improve their sleep and circadian rhythms. Each challenge lasts for 7 tracked nights, ranging from optimizing sleep habits to limiting caffeine intake, and more. Additional sleep improvement features embedded within the app include sleep sanctuary bedroom checks, sleep sounds, smart alarms, bedtime reminders, and sleep education blogs and science content.
  Other Names: SleepScore Mobile App; Dein Schlaf. Dein Tag. App
  Arms: Allocation to Sleep Improvement App

SUMMARY:
The study is a single-blinded randomized waitlist controlled trial that aims to assess changes in objective and self-report sleep improvement through use of a dynamic and personalized sleep improvement smartphone app and advice engine in those with poor sleep (i.e., subclinical threshold insomnia) when compared to a waitlist control group after 6 weeks and 12 weeks.

DETAILED DESCRIPTION:
Subclinical sleep dysfunction has a multitude of causes (e.g., environmental, cognitive, behavioral, or physiological) and symptoms (e.g., long sleep onset latency, short sleep duration, elevated wake after sleep onset and nighttime awakenings, poor sleep quality). A personalized and dynamic sleep improvement intervention tailored to an individual's lifestyle and specific needs may therefore be required to help nudge those with poor sleep towards sleep-promoting behaviors and attitudes. Digital and mobile health platforms are also highly scalable and cost-effective, thus allowing for widespread implementation across larger subclinical populations.

The purpose of the present study is to conduct a single-blinded randomized waitlist controlled trial to evaluate a novel smartphone application, Dein Schlaf. Dein Tag. powered by SleepScore, designed to both objectively measure and improve sleep. The Dein Schlaf. Dein Tag. app features a validated sonar sleep measurement tool and also provides dynamic and personalized sleep advice founded in the principles of cognitive behavioral psychology and sleep hygiene, offering a non-invasive and non-pharmacological behavioral intervention designed to improve sleep and circadian functioning in those with common sleeping difficulties. Participants will be randomly assigned to the sleep improvement app intervention or a waitlist control group. Online assessments on validated sleep and preventative health measures will take place at baseline, 6 weeks, and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* iOS user
* Sub-clinical threshold insomnia symptoms (Regensburg Insomnia Scale Score 13-24)
* ≥ 18 years old.
* Naive to the SleepScore Labs App
* Able to fully understand information on data protection and provide written informed consent

Exclusion Criteria:

* Non-iOS device users due to technical restrictions of the application
* Bedtime less than 6 hours
* Any of the following medical problems:

  * Untreated psychological disorder affecting sleep (e.g., depression, anxiety disorders, bipolar disorder, schizophrenia)
  * Current severe medical conditions (e.g. chronic pain, cancer)
* Any of the following medications/substance use:

  * Prescription sleep medications or regular use of over-the-counter sleep medications
  * Medication for other conditions (e.g., anxiety, ADHD) that affect sleep, e.g. antidepressants, antipsychotics
* Consumption of 3+ units of alcohol on 4 or more nights per week
* Recreational or nightly drug use
* Pregnant or nursing mothers
* Shift work
* Travel across 2 or more time zones during study period
* Sleeping more than 7 nights not at home during study period
* Users who newly received a diagnosis of a sleep disorders
* Users who start sleep or other psychoactive medication during the study period
* Use of other Sleep Tracking App's during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 637 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Schoebel, Prof, Principal Investigator — Ruhrlandklinik Essen
Locations (1):
- Ruhrlandklinik Essen, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD as data analysis will be conducted internally and raw IPD will not be shared with external researchers.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 754 individuals entered prescreening and/or expressed interest ('signed up'). After eligibility screening and completion of baseline, 637 participants were randomized and started: 318 to the app and 319 to waitlist. The difference (754 to 637) reflects screening processes and incomplete baseline assessments prior to randomization.
Groups:
- Allocation to Sleep Improvement App: Participants will be instructed to engage with the Dein Schlaf. Dein Tag. smartphone app, log their behaviors in-app, and track their sleep daily for the duration of the study (12 weeks). Participants will be instructed to start the sleep tracking device via their iOS device before lying down in bed and turning off the lights to go to sleep. In the morning, participants will turn off the sleep tracking device as soon as they wake up and decide to leave the bed. At the three time points (baseline, 6 weeks, and 12 weeks), participants will be instructed to complete online assessments on self-reported sleep quality, health perception, psychosocial factors and sleep-permissive behaviors (i.e., preventative health)
  Dein Schlaf. Dein Tag. sleep improvement application powered by SleepScore: The Dein Schlaf. Dein Tag. application powered by SleepScore is a validated sleep measurement application using sonar technology that also provides evidenced-based sleep advice and sleep education content based on a user's objectively measured nightly sleep data. As participants engage with the app, the Dein Schlaf. Dein Tag. application provides personalized and dynamic sleep content and sleep and circadian rhythm improvement advice based in the principles of sleep hygiene, sleep-circadian science, and cognitive behavioral psychology.
Period: Overall Study
Arm/Group | Allocation to Sleep Improvement App | Allocation to Waitlist Control Group
Started | 318 | 319
Completed | 194 | 285
Not Completed | 124 | 34
Not completed — Lost to Follow-up | 124 | 34

BASELINE CHARACTERISTICS:
Population: All randomized participants with non missing data
Groups:
- Total: Total of all reporting groups
Arm/Group | Allocation to Sleep Improvement App | Allocation to Waitlist Control Group | Total
Number analyzed (Participants) | 318 | 319 | 637
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (12) | 42 (13) | 42 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 242 | 253 | 495
  Male | 76 | 66 | 142
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 318 | 319 | 637

OUTCOME MEASURES:

1. Primary Outcome: Change in SF B Sleep Quality From Baseline to 6 Weeks
Description: SF B Sleep Quality (SQ): SF B (Görtelmeyer). Range 1-5; higher = better sleep quality.
Time Frame: Baseline and 6 weeks
Population: All randomized participants with non missing data at the specified follow up (intent to treat completer analysis). 6 week n: App 206; Control 286.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Allocation to Sleep Improvement App: Participants will be instructed to engage with the Dein Schlaf. Dein Tag. smartphone app, log their behaviors in-app, and track their sleep daily for the duration of the study (12 weeks). Participants will be instructed to start the sleep tracking device via their iOS device before lying down in bed and turning off the lights to go to sleep. In the morning, participants will turn off the sleep tracking device as soon as they wake up and decide to leave the bed. At the three time points (baseline, 6 weeks, and 12 weeks), participants will be instructed to complete online assessments on self-reported sleep quality, health perception, psychosocial factors and sleep-permissive behaviors (i.e., preventative health)
  Dein Schlaf. Dein Tag. sleep improvement application powered by SleepScore: The Dein Schlaf. Dein Tag. application powered by SleepScore is a validated sleep measurement application using sonar technology that also provides evidenced-based sleep advice and sleep education content based on a user's objectively measured nightly sleep data. As participants engage with the app, the Dein Schlaf. Dein Tag. application provides personalized and dynamic sleep content and sleep and circadian rhythm improvement advice based in the principles of sleep hygiene, sleep-circadian science, and cognitive behavioral psychology. Participants will also receive personalized sleep challenges tailored to improve their sleep and circadian rhythms.
Arm/Group | Allocation to Sleep Improvement App | Allocation to Waitlist Control Group
Number analyzed (Participants) | 206 | 286
score on a scale
  Baseline | 2.73 (0.51) | 2.73 (0.56)
  6-week follow-up | 2.98 (0.51) | 2.81 (0.60)
Statistical Analysis 1: Comparison: Allocation to Sleep Improvement App vs Allocation to Waitlist Control Group; Test type: Superiority; p < 0.0001, ANOVA; Repeated measures ANOVA (Group × Time; app vs control; baseline vs week 12)

2. Primary Outcome: Change in SF B Sleep Quality From Baseline to 12 Weeks
Description: SF B Sleep Quality (SQ): SF B (Görtelmeyer). Range 1-5; higher = better sleep quality.
Time Frame: Baseline and 12 weeks
Population: All randomized participants with non missing data at the specified follow up (intent to treat completer analysis). 12 week n: App 194; Control 285.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Allocation to Sleep Improvement App | Allocation to Waitlist Control Group
Number analyzed (Participants) | 194 | 285
score on a scale
  Baseline | 2.75 (0.50) | 2.73 (0.56)
  12-week follow-up | 3.05 (0.51) | 2.86 (0.64)
Statistical Analysis 1: Comparison: Allocation to Sleep Improvement App vs Allocation to Waitlist Control Group; Test type: Superiority; p = 0.0003, ANOVA; Repeated measures ANOVA (Group × Time; app vs control; baseline vs week 12)

3. Secondary Outcome: Changes in Overall Sleep Problems From Baseline to 6 Weeks
Description: PSQI Global Score: Range 0-21; higher = worse sleep quality; conventional cutoff >5 indicates poor sleep.
Time Frame: Baseline and 6 weeks
Population: Secondary analyses were conducted using an adherent to treatment approach, only including participants who did sufficiently engage with the app, that is, the subgroup of app users who tracked their sleep frequently (more than three times per week) between first activation and 6-week assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Allocation to Sleep Improvement App | Allocation to Waitlist Control Group
Number analyzed (Participants) | 121 | 286
score on a scale
  Baseline | 8.54 (3.02) | 8.47 (3.37)
  6-week follow-up | 7.14 (2.65) | 8.24 (3.57)
Statistical Analysis 1: Comparison: Allocation to Sleep Improvement App vs Allocation to Waitlist Control Group; Test type: Superiority; p = 0.0002, ANOVA; Repeated measures ANOVA (Group × Time; frequent app users vs control; baseline vs week 6)

4. Secondary Outcome: Changes in Feeling of Being Refreshed in the Morning From Baseline to 6 Weeks
Description: SF B Feeling Refreshed (GES): SF B GES subscale. Range 1-5; higher = better feeling of being refreshed.
Time Frame: Baseline and 6 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Allocation to Sleep Improvement App | Allocation to Waitlist Control Group
Number analyzed (Participants) | 121 | 286
score on a scale
  Baseline | 2.68 (0.63) | 2.68 (0.77)
  6-week follow-up | 2.86 (0.70) | 2.75 (0.78)
Statistical Analysis 1: Comparison: Allocation to Sleep Improvement App vs Allocation to Waitlist Control Group; Test type: Superiority; p = 0.0606, ANOVA; Repeated measures ANOVA (Group × Time; frequent app users vs control; baseline vs week 6)

5. Secondary Outcome: Changes in Health Measures From Baseline to 6 Weeks
Description: SF 12 (PCS & MCS): Norm based T scores (mean 50, SD 10); higher = better health status. We report PCS and MCS separately.
Time Frame: Baseline and 6 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Allocation to Sleep Improvement App | Allocation to Waitlist Control Group
Number analyzed (Participants) | 121 | 286
score on a scale
  Baseline physical wellbeing SF-12 | 52.70 (6.62) | 51.01 (8.76)
  6-week follow-up physical wellbeing SF-12 | 53.13 (8.09) | 50.45 (9.11)
  Baseline mental wellbeing SF-12 | 37.31 (6.15) | 38.16 (6.68)
  6-week follow-up mental wellbeing SF-12 | 38.56 (7.16) | 38.77 (6.69)
Statistical Analysis 1: Comparison: Allocation to Sleep Improvement App vs Allocation to Waitlist Control Group; SF-12 Physical Wellbeing; Test type: Superiority; p = 0.2056, ANOVA; Repeated measures ANOVA (Group × Time; frequent app users vs control; baseline vs week 6)
Statistical Analysis 2: Comparison: Allocation to Sleep Improvement App vs Allocation to Waitlist Control Group; SF-12 Mental Wellbeing; Test type: Superiority; p = 0.4186, ANOVA; Repeated measures ANOVA (Group × Time; frequent app users vs control; baseline vs week 6

6. Secondary Outcome: Changes in Mental Health Stress From Baseline to 6 Weeks
Description: PSS 10: 10 items scored 1-5; total 10-50; higher = more stress.
Time Frame: Baseline and 6 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Allocation to Sleep Improvement App | Allocation to Waitlist Control Group
Number analyzed (Participants) | 121 | 286
score on a scale
  Baseline | 28.62 (6.34) | 28.87 (6.35)
  6-week follow-up | 27.27 (6.97) | 28.62 (6.58)
Statistical Analysis 1: Comparison: Allocation to Sleep Improvement App vs Allocation to Waitlist Control Group; Test type: Superiority; p = 0.0754, ANOVA; Repeated measures ANOVA (Group × Time; frequent app users vs control; baseline vs week 6)

7. Secondary Outcome: Changes in Overall Sleep Problems From Baseline to 12 Weeks
Description: PSQI Global Score: Range 0-21; higher = worse sleep quality; conventional cutoff >5 indicates poor sleep.
Time Frame: Baseline and 12 weeks
Population: Secondary analyses were conducted using an adherent to treatment approach, only including participants who did sufficiently engage with the app, that is, the subgroup of app users who tracked their sleep frequently (more than three times per week) between first activation and 6-week assessment and completed the 12-week assessment; only those who continued frequent tracking until 12 weeks were included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Allocation to Sleep Improvement App | Allocation to Waitlist Control Group
Number analyzed (Participants) | 111 | 285
score on a scale
  Baseline | 8.50 (3.02) | 8.41 (3.35)
  12-week follow-up | 7.11 (2.77) | 7.88 (3.50)
Statistical Analysis 1: Comparison: Allocation to Sleep Improvement App vs Allocation to Waitlist Control Group; Test type: Superiority; p = 0.0137, ANOVA; Repeated measures ANOVA (Group × Time; frequent app vs control; baseline vs week 12)

8. Secondary Outcome: Changes in Feeling of Being Refreshed in the Morning From Baseline to 12 Weeks
Description: SF B Feeling Refreshed (GES): SF B GES subscale. Range 1-5; higher = better feeling of being refreshed.
Time Frame: Baseline and 12 weeks
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Allocation to Sleep Improvement App | Allocation to Waitlist Control Group
Number analyzed (Participants) | 111 | 285
score on a scale
  Baseline | 2.72 (0.63) | 2.67 (0.73)
  12-week follow-up | 2.98 (0.74) | 2.77 (0.78)
Statistical Analysis 1: Comparison: Allocation to Sleep Improvement App vs Allocation to Waitlist Control Group; Test type: Superiority; p = 0.0152, ANOVA; Repeated measures ANOVA (Group × Time; frequent app vs control; baseline vs week 12)

9. Secondary Outcome: Changes in Health Measures From Baseline to 12 Weeks
Description: as for outcome 5
Time Frame: Baseline and 12 weeks
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Allocation to Sleep Improvement App | Allocation to Waitlist Control Group
Number analyzed (Participants) | 111 | 285
score on a scale
  Baseline physical wellbeing SF-12 | 52.88 (6.59) | 51.22 (8.74)
  12-week follow-up physical wellbeing SF-12 | 53.08 (7.78) | 51.61 (8.75)
  Baseline mental wellbeing SF-12 | 37.80 (6.04) | 38.29 (6.61)
  12-week follow-up mental wellbeing SF-12 | 39.27 (6.53) | 38.19 (6.85)
Statistical Analysis 1: Comparison: Allocation to Sleep Improvement App vs Allocation to Waitlist Control Group; SF-12 Physical Wellbeing; Test type: Superiority; p = 0.8148, ANOVA; Repeated measures ANOVA (Group × Time; frequent app vs control; baseline vs week 12)
Statistical Analysis 2: Comparison: Allocation to Sleep Improvement App vs Allocation to Waitlist Control Group; SF-12 Mental Wellbeing; Test type: Superiority; p = 0.0523, ANOVA; Repeated measures ANOVA (Group × Time; frequent app vs control; baseline vs week 12)

10. Secondary Outcome: Changes in Mental Health Stress From Baseline to 12 Weeks
Description: PSS 10: 10 items scored 1-5; total 10-50; higher = more stress.
Time Frame: Baseline and 12 weeks
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Allocation to Sleep Improvement App | Allocation to Waitlist Control Group
Number analyzed (Participants) | 111 | 285
score on a scale
  Baseline | 28.05 (6.18) | 28.81 (6.40)
  12-week follow-up | 25.60 (6.57) | 27.48 (6.71)
Statistical Analysis 1: Comparison: Allocation to Sleep Improvement App vs Allocation to Waitlist Control Group; Test type: Superiority; p = 0.0729, ANOVA; Repeated measures ANOVA (Group × Time; frequent app vs control; baseline vs week 12)

ADVERSE EVENTS:
Time Frame: From randomization through 12 weeks of follow up.
Description: Non systematic assessment appropriate for a minimal risk behavioral/digital intervention. Participants were not systematically queried at each visit; however, any unanticipated problems or unexpected AEs would have been reported per protocol to the ethics committee. No deaths, serious AEs, or other AEs were reported during the randomized 12 week period.
Arm/Group | Allocation to Sleep Improvement App | Allocation to Waitlist Control Group
All-Cause Mortality (participants affected / at risk) | 0/318 | 0/319
Serious Adverse Events (participants affected / at risk) | 0/318 | 0/319
Other Adverse Events (participants affected / at risk) | 0/318 | 0/319

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-04-28): https://cdn.clinicaltrials.gov/large-docs/59/NCT05195359/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/59/NCT05195359/SAP_001.pdf